CLINICAL TRIAL: NCT05164796
Title: Intravascular Ultrasound Assessment of Coronary Artery at High Risk for Obstruction Following TAVI
Brief Title: IVUS Analysis for Coronary Obstruction in TAVI
Acronym: ICARO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Collaborators: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Flavio Ribichini, Professor, Universita di Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICARO
Record Dates: First submitted 2021-11-18; First posted 2021-12-21 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Occlusion
MeSH Terms: conditions — Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVUS-guided (Experimental)
  Interventions: Device: IVUS assessment of coronary ostia

INTERVENTIONS:
Device: IVUS assessment of coronary ostia — For coronary arteries at high-risk of obstruction during TAVI in native valves or valve-in-valve TAVI:
  * IVUS analysis before valve implantation (+ coronary angiogram) to detect any leaflet interference with the coronary ostium, existing prior to the transcatheter heart valve (THV) placement
  * IVUS analysis (+ coronary angiogram) after valve implantation in absence of acute coronary occlusion, to assess the patency of the ostium at-risk, the presence of native or degenerated surgical leaflet adjacent to the ostium, and the interaction of THV-frame with the coronary ostium.
  * In case of CHIMNEY stenting, re-assessment of the stent expansion and coronary ostia patency with IVUS.

SUMMARY:
Observational, prospective, single-arm and multi-center study to assess the safety and feasibility of IVUS imaging in the setting of TAVI and to describe the angiographic and intravascular ultrasound features in patients with coronary arteries deemed at high-risk for coronary artery obstruction following TAVI.

DETAILED DESCRIPTION:
CHIMNEY stenting is a reasonable strategy to manage catastrophic coronary artery obstruction (CAO). However, this technique is frequently used, not for acute catastrophic CAO (clinically evident), but preventively because the operator believes that CAO may occur on complete transcatheter heart valve (THV) deployment or after the protective coronary guidewire is withdrawn (3/5 of cases). Consequently, in current clinical practice, many patients receive CHIMNEY stents that are not required, and thus incur the associated risks of this procedure. To date, operators do not know how many patients, among those underwent preventive CHIMNEY, really required stenting, or on the contrary, did not. Also, accordingly, a real estimation of CAO incidence is not possible, but is likely higher than that reported in previous studies.

At present, no objective measures have been identified that could help operators decide when to deploy a CHIMNEY stent. If it could be demonstrated in the catheterization laboratory that the displaced native or bioprosthetic leaflets were sufficiently far away from the native coronary ostia and the risk for CAO was low, then unnecessary CHIMNEY stenting could be avoided.

Angiographic images do not provide sufficient information to clarify that. The investigation of a coronary ostium at risk of CAO from an intravascular point of view may reveal the presence of the displaced leaflet in front of them, or on the other hand, its absence, supporting operators in the decision to stent or not to stent.

In addition to the potential for IVUS to determine when CHIMNEY stenting should be used, this technique may also be used to optimize the results of CHIMNEY stenting when it has been deployed.

Moreover, IVUS can also be used to assess the result of the BASILICA technique after leaflet laceration.

The hypothesis is that the use of IVUS imaging for the assessment of patency of the coronary ostium and of the relationship of displaced valve leaflets towards the coronary arteries may reveal novel risk factors to predict which are not detectable by traditional angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Written informed consent
3. Diagnosis of symptomatic severe aortic stenosis, or clinically relevant degeneration of previously implanted surgical aortic valve bioprosthesis
4. Patient undergoing TAVI according to local institutional protocol and following Heart Team discussion.
5. High-quality ECG gated computed tomography (CT) scan of the heart and aorta
6. Presence of 2 or more of the following risk factors for CAO (high-risk):

6a. TAVI in native valves: height of the coronary ostium (<9 mm), sinuses of Valsalva width <30 mm, leaflet tips extending above the coronary ostia or the sino-tubular junction.

6b. VIV-TAVI (patients undergoing BASILICA as first prevention strategy are also included): surgical bioprosthesis type: with supra-annular position, high leaflet profile, externally mounted leaflets stented valve, stentless valves, and bulky leaflets, low-lying coronary ostia (< 9 mm from the ostia to the sewing ring), narrow sinuses of Valsalva (<30 mm by width for Valsalva sinuses), virtual THV-coronary (VTC) distance <4 mm, virtual THV-STJ (VT-STJ) distance < 2.5-3.5 mm: to be considered in cases where VTC >4mm but the leaflet extends above or very close (up to 2mm below) to the STJ plane.

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. Absence of informed consent
4. Angiographic or functional critical stenosis of the at-risk coronary artery (%DS > 70 for right coronary artery, > 50 for left main, or positive functional assessment), requiring revascularization regardless the risk of CAO.
5. Signs or symptoms of acute (unstable) myocardial ischemia
6. Reduced survival expectancy due to severe co-morbidities (<1 year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of IVUS assessement success | Within the same 1 procedural day
  Feasibility of IVUS assessement after the valve implantation (Yes, No)
Incidence of IVUS assessment-related adverse events | Within the same 1 procedural day
  Safety of IVUS assessement. Composite of any clinical complication related to the attempted insertion of the IVUS catheter into the coronary artery, including: dissection, perforation, thrombosis, or flow impairment of the at-risk coronary or damage to the aortic wall or the THV during insertion of the IVUS catheter prior to or after TAVI.

SECONDARY OUTCOMES:
CHIMNEY stenting rate | Within the same 1 procedural day
  Comparison between the actual rate of CHIMNEY stenting performed after the final IVUS assessment, and the rate of potential CHIMNEY stenting reported by operators on the only basis of CT and angiography images (before IVUS assessment). This will provide information about the number of stents that could be "spared" because deemed useless after the more accurate IVUS study
MACE | 1 month, 1 year.
  Major Adverse Cardiovascular Events (MACE) occurred among patients treated with CHIMNEY stenting or with a deferred stent strategy at discharge, 30-day and 1-year follow-up
IVUS-angiography agreement rate | Procedural 1 day
  The rate of agreement between angiography and IVUS evaluation of coronary ostia:
  1. rate of significant ostial stenosis as per angiography (%DS > 70 for RCA and > 50 for LM) vs IVUS assessment (lumen area < 4 mm2 for RCA and < 6 mm2 for LM).
  2. rate of leaflet footprint/floating mass detection by angiography vs IVUS
Stent-optimization rate | Procedural 1 day
  The rate of stent optimization (post-dilatation or adjunctive stents) guided by IVUS assessment (only in stented coronaries)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Ribichini, MD, Principal Investigator — Universita di Verona; Darren Mylotte, MD, PhD, Principal Investigator — National University of Ireland Galway, Ireland. University College Hospital Galway, Ireland.
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pighi M, Lunardi M, Pesarini G, Castriota F, Venturi G, Gottin L, Scarsini R, Ferrero V, Ribichini FL. Intravascular ultrasound assessment of coronary ostia following valve-in-valve transcatheter aortic valve implantation. EuroIntervention. 2021 Feb 19;16(14):1148-1151. doi: 10.4244/EIJ-D-20-00611. No abstract available. PMID 32894228